CLINICAL TRIAL: NCT01062828
Title: Defining Normal Citrulline Levels as a Diagnostic Tool for Screening of Gastrointestinal Disease in Premature Infants
Status: Terminated | Type: Observational
Why Stopped: Terminated: participants are no longer being enrolled
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Teresa del Moral, Associate professor, University of Miami
Other Study IDs: 20081180
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Premature Newborn; Necrotizing Enterocolitis
Keywords: Prematurity; Necrotizing Enterocolitis; Feeding Intolerance
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gestational age < 32 weeks: Premature infants with gestational age between <32 weeks regardless of birth weight
  Interventions: Diagnostic Test: Citrulline samples

INTERVENTIONS:
Diagnostic Test: Citrulline samples — Citrulline samples will be collected at the time of other lab work twice a week from enrollment until 40 weeks postconceptional age and once a week until 44 weeks postconceptional age (1 month corrected age) OR discharge from NICU(whichever is soonest). In subgroup developing NEC, citrulline samples will be collected twice a week from enrollment until discharge from NICU or death.

SUMMARY:
Since the first description of citrulline as a potential marker for intestinal function in 1998, its use has been investigated in a variety of disease processes including Short Bowel Syndrome, Celiac disease, chemotherapy and radiation induced intestinal injury, infections producing intestinal cytopathic effects like Adenovirus, and predicting rejection in intestinal transplantation. The use of citrulline levels as a diagnostic tool to predict gastrointestinal disease in the premature population has not been properly addressed.

The introduction of enteral nutrition in the premature infant is a process of trial and error, knowing that the immaturity of the gastrointestinal system may lead to frequent episodes of feeding intolerance. This is augmented by the fear of the development of necrotizing enterocolitis (NEC) once feeds are commenced. NEC is a condition characterized by disruption of the intestinal epithelial barrier, a pathogenic process shared with some of the conditions mentioned above for which citrulline has proven clinically useful.

A normal pattern of citrulline production has not been established in the premature population. Previous studies have shown decreased levels of glutamine and arginine in premature infants up to 10 days prior to the development of necrotizing enterocolitis. Glutamine and arginine are two amino acids closely involved in the synthesis and catabolism of citrulline.

The investigators therefore hypothesize that defining a normal pattern of citrulline production in the premature population may prove to be a clinically useful diagnostic tool to screen for gastrointestinal disease.

DETAILED DESCRIPTION:
The use of citrulline levels as a diagnostic tool to predict gastrointestinal disease in the premature population has not been properly addressed.

ELIGIBILITY:
Inclusion Criteria:

1. Premature infants with gestational age between <32 weeks regardless of birth weight

Exclusion Criteria:

1. Inborn errors of metabolism
2. Need for exchange transfusion
3. Multiple congenital anomalies
4. Renal failure (defined as urine output <1ml/k/h >24h, creatinine >1.8, or diagnosis of "non-oliguric renal failure" as determined by Pediatric nephrology)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Premature infants with gestational age between <32 weeks regardless of birth weight born at University of Miami/Holtz Children's Hospital Neonatal Intensive Care Unit, or transferred in within the first 72h of life.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to establish the normal pattern of citrulline concentration in the premature population, infants born <32 weeks gestation, which represents normal maturity of the intestinal glutamine pathway. | From birth to one month corrected age (Gestational age 44 weeks) or discharge from neonatal intensive care unit (NICU)
  Levels of citrulline concentration in premature infants

SECONDARY OUTCOMES:
A secondary outcome, in the subgroup of infants who develop necrotizing enterocolitis, will be to evaluate the pattern of citrulline concentration prior to its development. | From birth until discharge from NICU
  levels of citrulline concentration in prematureinfants with NEC

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Garcia, MD, Study Director — University of Miami, Dept of Pediatrics, Division of GI, Hepatology and Nutrition; Teresa Del Moral, MD, Principal Investigator — University of Miami, Dept of Pediatrics, Division of Neonatology; John Thompson, MD, Study Chair — The Children's Hospital at Montefiore
Locations (1):
- Holtz Children's Hospital- University of Miami/Jackson Memorial Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No